CLINICAL TRIAL: NCT03782259
Title: Effects of SGLT-2 Inhibition With Dapagliflozin on Myocardial Fibrosis and Inflammation as Assessed by Cardiac MRI With T1- and T2-mapping in Patients With Type-2 Diabetes
Brief Title: Effects of SGLT-2 Inhibition on Myocardial Fibrosis and Inflammation as Assessed by Cardiac MRI in Patients With DM2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Francis Kim, Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: STUDY00004982; ESR 17-13124 (Other: AstraZeneca Pharmaceuticals, LP)
Record Dates: First submitted 2018-10-24; First posted 2018-12-20 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Mellitus; Myocardial Fibrosis; Myocardial Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocarditis | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind and placebo controlled cardiac MRI study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 10mg tabs placebo matching dapagliflozin.
  Interventions: Other: Placebo
- Active (Active Comparator): 10mg tabs of dapagliflozin
  Interventions: Drug: dapagliflozin

INTERVENTIONS:
Drug: dapagliflozin — Subjects will either receive 10mg tabs of dapagliflozin or identical looking placebo - inactive medication. Subjects have an equal chance of receiving dapagliflozin or placebo. Which treatment subjects receive is decided at random by a computer (purely by chance, like the tossing of a coin). Neither subjects nor the Study Site personnel will know which treatment subjects are assigned to. The study drug must be taken daily. The subject's other medications will not be changed by the study.
  Other Names: Forxiga
  Arms: Active
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
There is an unmet need for Cardiovascular Disease (CVD) risk reduction in patients with Type 2 Diabetes. In recent trials there has been promising findings of more effective glucose management and reductions in overall CVD events and hospitalization for heart failure with SGLT-2 inhibition. Using the capability of cardiac MRI with T1- and T2-mapping in assessments of myocardial fibrosis and inflammation, the investigators propose to conduct a clinical trial to investigate the effects of SGLT-2 inhibition with dapagliflozin on myocardial strain, fibrosis and inflammation as assessed by cardiac MRI with T1- and T2-mapping in patients with type-2 diabetes.

Over approximately 12 months subjects will have 6 clinical visits at the investigators research clinic. During this time subjects will be randomized to receive either active 10mg dapagliflozin or a matching placebo. 2 MRI scans at one of the two University of Washington research imaging centers will take place. One at randomization and the second scan will occur approximately 12 months after the first scan.

DETAILED DESCRIPTION:
Given the unmet needs for CVD risk reduction in patients with Type 2 Diabetes Mellitus (T2DM), the promising findings of more effective glucose management and reductions in overall CVD events and hospitalization for heart failure with SGLT-2 inhibition demonstrated in recent trials, and the capability of cardiac MRI (CMRI) with T1- and T2-mapping in assessments of myocardial fibrosis and inflammation, the investigators propose to conduct a staged research program using adaptive study design to investigate the effects of SGLT-2 inhibition with dapagliflozin on myocardial strain, fibrosis and inflammation as assessed by cardiac MRI with T1- and T2-mapping in patients with type-2 diabetes.

A total of 60 subjects with >=18 years of age, type-2 diabetes history >=5 years and HbA1C 7-10% will be randomized at 1:1 to Dapagliflozin 10mg or matching placebo once daily for 1 year. All subjects will be followed every 3 months for clinical and laboratory evaluations and assessments. All subjects will undergo CMRI at baseline and 1 year.

The primary myocardial strain endpoint includes global myocardial longitudinal strain (GLS). Myocardial fibrosis endpoint is change in extracellular volume fraction (ECV) as assessed by T1-mapping over 12 months. ECV combines native and contrast-enhanced T1 mapping. The change of the T1 relaxation rate (i.e., 1/T1) in blood between pre- and post-contrast imaging is converted with the blood hematocrit into a reference for plasma T1, which serves as reference for the T1 changes in tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 18 years of age
2. Subjects with type-2 diabetes history >=5 years
3. HbA1C 7-10% with glucose control medications including insulin, metformin or sulfonylurea
4. Medically stable
5. Willing to participate and sign informed consent.

Exclusion Criteria:

1. Contraindication to MRI
2. Currently or within last three months treatment with a SGLT2 inhibitor
3. Currently taking glucagon-like peptide (GLP)-1 receptor antagonist
4. Glomerular filtration rate (GFR) <60 mL/min/1.73 m2
5. Unstable or rapidly progressive renal disease
6. Hypotension with systolic blood pressure (SBP) <100 mmHg
7. Hypersensitivity to dapagliflozin or any excipients
8. Patients with severe hepatic impairment (Child-Pugh class C)
9. Patients with active hepatitis B or C infection
10. Any of the following CV/Vascular Diseases within 3 months prior to signing the consent at enrollment, as assessed by the investigator:

    1. Myocardial infarction
    2. Cardiac surgery or revascularization (CABG/PTCA)
    3. Unstable angina
    4. Heart Failure - New York Heart Association (NYHA) Class IV
    5. Transient ischemic attack (TIA) or significant cerebrovascular disease
    6. Unstable or previously undiagnosed arrhythmia
    7. Established peripheral artery disease (PAD)

(18) Active bladder cancer (19) Recent episode of Diabetic ketoacidosis (DKA), frequent episodes of DKA (20) High risk of fractures, amputations and fibrosis (21) Women of child-bearing potential (ie, those who are not chemically or surgically sterilized or who are not post-menopausal) who have a positive pregnancy test at enrollment or randomization, OR women who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator, from the time of signing the informed consent until two weeks after the last dose of study drug, OR women who are breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Qiao Zhao, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Naumova AV, Cunha GM, Kim NJ, Lu J, Isquith D, Chu B, Maynard C, Mahdavi A, Firoozeh N, Ordovas K, Zhao XQ, Kim F. Dapagliflozin-Associated Reduction in Liver Fat Is Independent of Weight Loss in Patients With Type 2 Diabetes. Obesity (Silver Spring). 2026 Feb 2. doi: 10.1002/oby.70134. Online ahead of print. PMID 41629250
- [Derived] Wang DD, Naumova AV, Isquith D, Sapp J, Huynh KA, Tucker I, Balu N, Voronyuk A, Chu B, Ordovas K, Maynard C, Tian R, Zhao XQ, Kim F. Dapagliflozin reduces systemic inflammation in patients with type 2 diabetes without known heart failure. Cardiovasc Diabetol. 2024 Jun 7;23(1):197. doi: 10.1186/s12933-024-02294-z. PMID 38849829
- [Derived] Wang D, Naumova A, Isquith D, Sapp J, Huynh KA, Tucker I, Balu N, Voronyuk A, Chu B, Ordovas K, Maynard C, Tian R, Zhao XQ, Kim F. Dapagliflozin Reduces Systemic Inflammation in Patients with Type 2 Diabetes Without Known Heart Failure. Res Sq [Preprint]. 2024 Mar 25:rs.3.rs-4132581. doi: 10.21203/rs.3.rs-4132581/v1. PMID 38585865

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin: 10mg tabs of dapagliflozin
  dapagliflozin: Subjects will either receive 10mg tabs of dapagliflozin or identical looking placebo - inactive medication. Subjects have an equal chance of receiving dapagliflozin or placebo. Which treatment subjects receive is decided at random by a computer (purely by chance, like the tossing of a coin). Neither subjects nor the Study Site personnel will know which treatment subjects are assigned to. The study drug must be taken daily. The subject's other medications will not be changed by the study.
Period: Overall Study
Arm/Group | Placebo | Dapagliflozin
Started | 31 | 31
Completed | 29 | 27
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Moved out of state | 0 | 2
Not completed — MRI incompatibility: Pacemaker implanted prior to subject final MRI scan | 0 | 1
Not completed — Subject discontinued intervention | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11) | 62 (9) | 62 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 27 | 30 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 20 | 23 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62
Hypertension [Count of Participants; unit: Participants] | 19 | 19 | 38
Diabetes mellitus [Count of Participants; unit: Participants] | 31 | 31 | 62
Hyperlipidemia [Count of Participants; unit: Participants] | 18 | 21 | 39
Current smoker [Count of Participants; unit: Participants] | 3 | 2 | 5
Family history myocardial infarction [Count of Participants; unit: Participants] | 11 | 12 | 23
Family history stroke [Count of Participants; unit: Participants] | 11 | 14 | 25
History myocardial infarction [Count of Participants; unit: Participants] | 2 | 1 | 3
Angina [Count of Participants; unit: Participants] | 2 | 1 | 3
Coronary artery bypass surgery [Count of Participants; unit: Participants] | 2 | 0 | 2
Percutaneous coronary intervention [Count of Participants; unit: Participants] | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Extracellular Volume Fraction (ECV)
Description: Cardiac MRI using T1-mapping is capable of quantifying myocardial extracellular volume (ECV), a surrogate of fibrosis, with excellent inter- and intra-observer variability. Cardiac fibrosis was assessed by cardiac MRI T1 mapping to calculate ECV at two timepoints, baseline and at approximately 1 year. ECV combines native and contrast-enhanced T1 mapping.
  Extracellular Volume (ECV) maps were generated offline using MATLAB software. ECV was calculated from native and post-contrast T1 values for blood and myocardial tissue, the partition coefficient lambda (λ), and hematocrit using the following formulas: ECV = λ(1-hematocrit); λ = (1/T1 myocardium post-contrast-1/T1 myocardium-native)/(1/T1 blood post-contrast-1/T1 blood-native).
Time Frame: Approximately 12 Months
Measure: Mean (Standard Deviation); unit: Percentage of total tissue volume
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 29 | 27
Percentage of total tissue volume
  Baseline | 28.5 (2.1) | 27.7 (2.9)
  1 year | 28.7 (2.3) | 28.4 (2.0)
  Difference (1 year - baseline) | 0.24 (2.16) | 0.71 (2.75)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; Test type: Superiority; p < 0 .0125, Wilcoxon (Mann-Whitney) — Given that there were 4 separate comparisons of the primary outcomes, the level of significance was adjusted from 0.05 to 0.0125 (.05/4) using the Bonferroni correction; There were no adjustments for covariates

2. Primary Outcome: Global Myocardial Strain
Description: Global myocardial strain measured from cardiac MRI with T1-mapping at two timepoints. MRI at Randomization and MRI at approximately 12 Months. Myocardial strain measurements with feature tracking will be performed to measure myocardial strain from the Balanced Steady State Free Precession (bSSFP) short-axis and long-axis cine images. Long-axis cine images will be further used to compute global myocardial strain. Ancova test with adjusted for baseline global myocardial strain will be used to compare change in global myocardial strain over 12 months between 2 treatment groups.
  Global myocardial strain reported as longitudinal, radial, and circumferential at baseline and 1 year.
Time Frame: Approximately 12 Months
Measure: Mean (Standard Deviation); unit: Change in length as a percentage
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 31 | 31
Change in length as a percentage
  Global myocardial longitudinal strain - Baseline | -11.0 (3.9) | -12.9 (3.4)
  Global myocardial longitudinal strain - 1 year | -11.3 (5.1) | -12.0 (3.8)
  Global myocardial longitudinal strain - Difference (1 year - baseline) | -0.24 (5.32) | 0.88 (4.06)
  Global myocardial radial strain - Baseline | 27.3 (7.1) | 31.2 (8.7)
  Global myocardial radial strain - 1 year | 31.3 (10.4) | 33.9 (9.5)
  Global myocardial radial strain - Difference (1 year - baseline) | 4.01 (10.19) | 2.71 (9.38)
  Global myocardial circumferential strain - Baseline | -15.7 (2.8) | -17.8 (2.9)
  Global myocardial circumferential strain - 1 year | -16.7 (2.9) | -17.7 (3.6)
  Global myocardial circumferential strain - Difference (1 year - baseline) | -0.97 (3.28) | 0.05 (3.21)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; Test type: Superiority; p < 0 .0125, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; There were no adjustments for covariates

3. Secondary Outcome: T2 Relaxation Time
Description: Change from baseline in T2 relaxation time measured from cardiac MRI with T2-mapping at two timepoints. MRI at Randomization and MRI at approximately 12 Months
Time Frame: Approximately 12 Months
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Active
Number analyzed (Participants) | 31 | 31
milliseconds
  Baseline | 48.6 (3.3) | 50.5 (4.3)
  1 year | 50.2 (3.8) | 50.0 (5.7)
  Difference (1 year - baseline) | 1.61 (4.14) | -0.51 (6.59)

4. Other Pre Specified Outcome: Fasting Glucose
Description: Fasting glucose assessed at Baseline and every 3 months for approximately 12 months, Baseline and 12 months reported
Time Frame: Approximately 12 Months
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 31 | 31
mg/dL
  Baseline | 164.5 (46.4) | 159.8 (42.5)
  1 year | 161.0 (55.9) | 126.8 (36.9)
  Difference (1 year - baseline) | -3.48 (39.56) | -33.04 (55.08)

5. Other Pre Specified Outcome: HbA1C
Description: Hemoglobin A1c (HbA1c) assessed at Baseline and every 3 months for approximately 12 months, Baseline and 12 months reported
Time Frame: Approximately 12 Months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 31 | 31
percentage
  Baseline | 7.8 (0.9) | 7.9 (.8)
  1 year | 8.0 (1.0) | 7.4 (.8)
  Difference (1 year - baseline) | 0.11 (1.17) | -.52 (0.95)

6. Other Pre Specified Outcome: hsCRP
Description: Inflammatory marker hsCRP assessed at Baseline and every 6 months for approximately 12 months, Baseline and 12 months reported
Time Frame: Approximately 12 Months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 31 | 31
mg/dL
  Baseline | 2.4 (.5) | 1.7 (1.6)
  1 year | 1.8 (.3) | 2.5 (4.1)
  Difference (1 year - baseline) | .12 (2.20) | 0.81 (2.95)

ADVERSE EVENTS:
Time Frame: Study screening visit to subject completion, approximately 13 months per subject.
Description: Adverse events were assessed at each of the subject visits.
Arm/Group | Placebo | Active
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Active (N=31)
Non-ST-elevation myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — PI determined not related to study intervention with causality as pre-existing/underlying disease - ASCVD, Diabetes.

LIMITATIONS AND CAVEATS:
* Relatively small trial was not powered to detect small effect sizes.
* Animal studies of SGLT2 inhibition used direct pathologic examination of inflammation and fibrosis; Cardiac MRI is known to be less sensitive.
* 12-month treatment may not have been sufficient to detect meaningful changes in inflammation, fibrosis, and strain.
* No matched, non-diabetic control group.
* Higher ECV values (>32) are associated with worse outcomes with known myocarditis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT03782259/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03782259/ICF_001.pdf